CLINICAL TRIAL: NCT04637087
Title: Precision Medicine in Ischemic Stroke and Atrial Fibrillation
Acronym: PreMISe-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Christopher D. Anderson, MD, MMSc, Division Chief, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020P001382
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Ischemic Stroke
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atrial Fibrillation Risk Estimation Tool (Experimental): For eligible patients presenting with an acute ischemic stroke, a clinical atrial fibrillation risk estimation tool will be displayed in the patient's electronic health record through a best practice alert (BPA). The alert will display for the stroke neurologist caring for the patient when they first open the patient's chart. The neurologist may accept the automatically generated atrial fibrillation risk score displayed in the BPA, may modify some of the inputs of the score based on the patient's personal medical history and re-calculate, or may choose to dismiss the BPA.
  Interventions: Other: Atrial fibrillation risk electronic health record alert

INTERVENTIONS:
Other: Atrial fibrillation risk electronic health record alert — Electronic health record best practice alert which displays patient's 5-year risk of developing atrial fibrillation

SUMMARY:
The overall goal of this study is to minimize morbidity due to Atrial Fibrillation (AF). The specific objective is to develop and implement a rational and personalized approach to AF risk estimation that can inform management decisions with ischemic stroke. The investigators propose to develop a clinical AF risk estimation tool in the electronic health record and to test the effectiveness of implementing a clinical AF risk estimation tool into care for use by stroke neurologists during the care of acute ischemic stroke patients at Massachusetts General Hospital. The investigators will evaluate cardiac monitoring utilization calibrated to AF risk by stroke neurologists using a custom electronic health record (EHR) notification module.

The investigators hypothesize that cardiac rhythm monitoring utilization will be positively correlated with the predicted risk of AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Presenting with a primary diagnosis of ischemic stroke or transient ischemic attack admitted to Massachusetts General Hospital inpatient stroke service

Exclusion Criteria:

* Patients not meeting above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac rhythm monitoring | 6-months
  Incidence of any cardiac rhythm monitoring in the 6-month follow-up period following discharge for an acute ischemic stroke. Cardiac rhythm monitoring will be ascertained based on electronic health record documentation.

SECONDARY OUTCOMES:
Proportion of patients with implantable loop recorder orders | 12-months
  Proportion of patients with implantable loop recorder ordered at discharge, 6-months, and 12-months. Implantable loop recorder orders will be ascertained based on electronic health record documentation.
Proportion of patients with ambulatory wearable cardiac rhythm monitoring orders | 12-months
  Proportion of patients with wearable cardiac rhythm monitor ordered at discharge, 6-months, and 12-months. Wearable cardiac rhythm monitoring orders will be ascertained based on electronic health record documentation.
Proportion of patients with cardiac monitor ordered by neurologist | 1-month
  Proportion of patients with cardiac monitor ordered by the neurologist at discharge. Cardiac monitor orders by the neurologist will be ascertained based on electronic health record documentation.
Proportion of patients with a new atrial fibrillation diagnosis | 12-months
  Proportion of patients with a new diagnosis of atrial fibrillation at 12-months following discharge for acute ischemic stroke based on electronic health record documentation.
Proportion of patients with recurrent stroke | 12-months
  Proportion of patients with recurrent stroke occurring within 12-months of discharge for an initial acute ischemic stroke. Recurrent stroke will be ascertained based on electronic health record documentation.
Proportion of patients deceased | 12-months
  Proportion of patients who die within 12-months of discharge for acute ischemic stroke. Death will be ascertained based on electroni health record documentation.
Proportion of patients with transesophageal echocardiogram utilization | 3-months
  Proportion of patients with transesophageal echocardiogram (TEE) within 3-months of discharge for acute ischemic stroke. Transesophageal echocardiogram utilization will be ascertained based on electronic health record documentation.
Proportion of patients with oral anticoagulation prescription | 12-months
  Proportion of patients with a new prescription for oral anticoagulation within 12-months of discharge following acute ischemic stroke. Prescriptions for oral anticoagulation will be ascertained based on electronic health record documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Anderson, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ashburner JM, Tack RWP, Khurshid S, Turner AC, Atlas SJ, Singer DE, Ellinor PT, Benjamin EJ, Trinquart L, Lubitz SA, Anderson CD. Impact of a clinical atrial fibrillation risk estimation tool on cardiac rhythm monitor utilization following acute ischemic stroke: A prepost clinical trial. Am Heart J. 2025 Jun;284:57-66. doi: 10.1016/j.ahj.2025.02.010. Epub 2025 Feb 18. PMID 39978665